CLINICAL TRIAL: NCT07205120
Title: Fluid Guided Heart Failure Treatment
Brief Title: Fluid Guided Heart Failure Treatment at the Cleveland Clinic
Acronym: FIGHT-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bodyport Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-529
Record Dates: First submitted 2025-09-24; First posted 2025-10-03 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
Keywords: scale
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Interventional arm (Experimental): Participants will begin receiving fluid-guided care when they begin using the device in the outpatient (home) setting.
  Participants will be monitored per routine clinical care and receive study follow-up visits at 45- and 90-days to assess clinical status, events, and medication changes.
  Interventions: Device: Heart Failure Management Intervention

INTERVENTIONS:
Device: Heart Failure Management Intervention — Participants will receive access to their weight and fluid levels on the Cardiac Scale and through the Bodyport Patient Portal. The provider will receive access to the Congestion Index, alerts, and Clinical Dashboard to support the remote management of the participant. The provider will receive a notice when an alert is generated and twice weekly reminders until the Congestion Index returns below an alert threshold. When an alert is generated, providers will attempt to contact the participant and will be encouraged to follow the recommendations contained within the ARG. Providers will also be encouraged to provide feedback and suggest improvements to the ARG throughout the study. Any changes to medical therapy resulting from an alert will be documented in the Bodyport Clinical Dashboard.

SUMMARY:
FIGHT-HF is an exploratory non-randomized open-label study evaluating a heart failure management intervention.

The goal of this pilot is to assess the performance of a fluid-guided heart failure management program and Alert Response Guide (ARG) using the Bodyport Cardiac Scale and Congestion Index in 50 adult participants with acute and chronic heart failure, who are followed by a Cleveland Clinic cardiologist.

DETAILED DESCRIPTION:
This study will assess the clinical integration of the Cardiac Scale and a composite biomarker algorithm, the Congestion Index and Alert, into existing health system workflows for HF management. The data collected in this study will be used to test and refine existing Congestion Index-guided HF management protocols contained within an Alert Response Guide (ARG). The final Alert Response Guide may be further validated in future randomized control trials.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for acute decompensated heart failure
* Age 21 years or older
* Able to speak and read English

Exclusion Criteria:

* New York Heart Association functional class IV symptoms
* Received or are scheduled to receive a heart transplant or ventricular assist - device in the next 12 months
* Have a glomerular filtration rate of less than 25 mL/min while nonresponsive to diuretic therapy or on chronic renal dialysis
* Have a history of regularly scheduled intravenous HF therapy (e.g., inotropes or diuretics)
* Have a life expectancy of less than 12 months
* Are pregnant or plan to become pregnant during the next 12 months
* Weigh greater than 375 lbs
* Unable to stand on two bare feet without assistance

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Congestion Index Alert Statistics | From enrollment to the end of the study duration at 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No